CLINICAL TRIAL: NCT04594629
Title: Efficacy of Nebulized PGI2 Versus Nebulized Nitroglycerine for Management of Pulmonary Hypertension After Valve Replacement Surgeries
Brief Title: PGI2 Versus Nitroglycerine for Management of Pulmonary Hypertension After Valve Surgeries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Assistant professor of Anaesthesiology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 70/2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Hypertension
Keywords: PGI2; Nitroglycerine; valve replacement surgery; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nitroglycerine group (Sham Comparator): Patients of nitroglycerine group received nebulized nitro glycerine (a vial contains 50 mg nitroclycerine ), its starting concentration was 200 mcg/ml with nitro glycerine was delivered at 2.5-5 mcg/kg/min (5 mg, 1 mg/ml) over 10 minutes by ultrasonic nebuliser connected to the inspiratory limb of the breathing circuit
  Interventions: Drug: Nitroglycerin
- PGI2 group (Active Comparator): Patients of PGI2 group received nebulized PGI2 (epoprostenol), 20000 ng/ml (Flolan; Glaxo Wellcome Inc, Research Triangle Park, NC) (60 ml syringe of PGI2 with concentration 20000 ng/ml was attached to an intravenous pump which delivers a titrating rate of 8 ml/h to the nebulizer compartment (MiniHEART nebulizer; Westmed, Tucson, Ariz) fixed to the inspiratory limb of the breathing circuit or to the face mask with venturi accessory for sprinkling. The nebulizer was filled with 15 ml PGI2 with nebulized oxygen flow rate 3 litres.
  Interventions: Drug: PGI2

INTERVENTIONS:
Drug: Nitroglycerin — Patients of nitroglycerine group received nebulized nitro glycerine (a vial contains 50 mg nitroclycerine ), its starting concentration was 200 mcg/ml with nitro glycerine was delivered at 2.5-5 mcg/kg/min (5 mg, 1 mg/ml) over 10 minutes by ultrasonic nebuliser connected to the inspiratory limb of the breathing circuit
  Other Names: N group
  Arms: nitroglycerine group
Drug: PGI2 — Patients of PGI2 group received nebulized PGI2 (epoprostenol), 20000 ng/ml (Flolan; Glaxo Wellcome Inc, Research Triangle Park, NC) (60 ml syringe of PGI2 with concentration 20000 ng/ml was attached to an intravenous pump which delivers a titrating rate of 8 ml/h to the nebulizer compartment (MiniHEART nebulizer; Westmed, Tucson, Ariz) fixed to the inspiratory limb of the breathing circuit or to the face mask with venturi accessory for sprinkling. The nebulizer was filled with 15 ml PGI2 with nebulized oxygen flow rate 3 litres
  Other Names: PG group
  Arms: PGI2 group

SUMMARY:
This study was conducted in 120 patients aged from 54-65 years scheduled for elective valve replacement surgeries. Patients were randomly allocated to nitro glycerine or PGI2 groups. Patients of nitro glycerine group received nebulized nitro glycerine at a rate of 2.5-5 mcg/kg/min (5 mg, 1 mg/ml) over 10 minutes by ultrasonic nebuliser. Patients of PGI2 group received nebulized PGI2 (epoprostenol), 20000 ng/ml (20000 ng/ml in 60 ml syringe was attached to an intravenous pump which delivers a titrating rate of 8 ml/h . The primary outcome was mean pulmonary artery pressure. The secondary outcomes included mean arterial blood pressure (MAP) (mmHg), PaO2/FiO2 ratio, cardiac index (CI) (l/min/m2) right ventricular ejection fraction (RVEF), central venous pressure(CVP) , 30-day mortality rate and the incidence of complications such as facial flushing, hypotension and re-exploration for bleeding.

DETAILED DESCRIPTION:
Postoperative pulmonary hypertension (PHT) is the most challenging complication of valvular heart disease about 73% of the patients particularly in those posted for mitral valve replacement surgery Methods This prospective study was conducted in 120 patients aged from 54-65 years scheduled for elective valve replacement surgeries. Patients were randomly allocated to either nitro glycerine or PGI2 groups. Patients of nitro glycerine group received nebulized nitro glycerine (its starting concentration was 200 mcg/ml); nitro glycerine was delivered at a rate of 2.5-5 mcg/kg/min (5 mg, 1 mg/ml) over 10 minutes by ultrasonic nebuliser connected to the inspiratory limb of the breathing circuit. Patients of PGI2 group received nebulized PGI2 (epoprostenol), 20000 ng/ml (20000 ng/ml in 60 ml syringe was attached to an intravenous pump which delivers a titrating rate of 8 ml/h to the nebulizer compartment. The primary outcome was mean pulmonary artery pressure. The secondary outcomes included mean arterial blood pressure (MAP) (mmHg), PaO2/FiO2 ratio, cardiac index (CI) (l/min/m2) right ventricular ejection fraction (RVEF), central venous pressure(CVP) measured at the end of cardiopulmonary bypass then 30 minutes after start of treatment then 4 hours after start of treatment, 30-day mortality rate and the incidence of complications such as facial flushing, hypotension and re-exploration for bleeding.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 66 years old
* elective valve replacement surgery
* pulmonary arterial hypertension

Exclusion Criteria:

* Emergency surgery
* severe renal and hepatic dysfunction
* uncontrolled supraventricular arrhythmia
* those requiring preoperative inotropes

Ages: 54 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
mean pulmonary artery pressure | baseline, 30 minutes after start of study drug, 4 hours after start of study drug
  decrease of mean pulmonary artery pressure

SECONDARY OUTCOMES:
mortality | 30 days postoperative
  rate of mortality
central venous pressure | at the end of cardiopulmonary bypass (baseline values) then 30 minutes after start of treatment then 4 hours after start of treatment
  measurement of central venous pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Shoeb, Study Director — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol, SAP
Time Frame: 5-6 months
Access Criteria: The collected data are coded, tabulated, and statistically analyzed using statistical package for social sciences software, version 17.0 (SPSS Inc., Chicago, Illinois, USA). Descriptive statistics are carried out for numerical parametric data and presented as mean±SD, whereas categorical data are presented as number and percentage. Variables such as demographic data and comorbidities are compared using the χ2-test. A P value less than 0.05 was considered significant.